CLINICAL TRIAL: NCT06769646
Title: SPRING - Assess the Clinical Care Pathway of Population With T2D and CKD in Four European Countries Using Real-world Data
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8385; U1111-1313-1011 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-12-09; First posted 2025-01-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus (T2D) and Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with T2D in THIN databases: Individuals from the THIN® France, THIN® Italy, THIN® Spain and THIN® UK databases living with T2D and CKD
  Interventions: Other: No tretament given

INTERVENTIONS:
Other: No tretament given — No treatment given

SUMMARY:
This study is being carried out in 4 countries (France, Italy, Spain and the UK) to understand the clinical care pathway of population living with type 2 diabetes who also have evidence of chronic kidney disease.

The primary objective is to describe the population with T2D and CKD in terms of demography, clinical characteristics and medication use by CKD stage.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years old or older) diagnosed with T2D and treated with an antidiabetic medication before or at index date, set up on 1 January 2021
2. With evidence of Kidney damage before or at index date:

   1. diagnosed with CKD
   2. or with a record of eGFR below 60 ml/min/1.73 m^2
   3. or with a record of uACR above 30 mg/g
3. Consulting a GP (all countries) or an Endocrinologist (France, Spain, Italy) or a Nephrologist (Spain) of the THIN® network.

Exclusion Criteria:

1. aged less than 18 years old at index date
2. less than 360 days prior index date
3. less than 360 days after index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals from the THIN® France, THIN® Italy, THIN® Spain and THIN® UK databases living with T2D and CKD
Sampling Method: Probability Sample
Enrollment: 110074 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of various CKD stages among patients with type 2 diabetes in the THIN database | From the registration date to 1 January 2021
  * Distribution of CKD stages, as determined by eGFR, in patients with and w/out CKD diagnosis
  * (+/- ACD-10 code for CKD) in cohort of patients diagnosed with T2D.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational site, Bangalore, India

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com